CLINICAL TRIAL: NCT02736903
Title: Efficacy of Mobile-based Online Social Network Intervention to Increase Physical Activity Among Young African American Women
Brief Title: Mobile-based Online Social Network Intervention to Increase Physical Activity
Acronym: PennFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 823881
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual intervention (Active Comparator): Behavioral: PennFit mobile individual intervention. Participants were given a Fitbit (zip) to track their daily exercises. Participants used the PennFit app to track their own daily steps and the minutes for vigorous, moderate, and muscle-strengthening exercises that they completed for each day. Participants also received system-generated notifications that reminded them to wear their Fitbit in the morning and to log their activity minutes in the evening.
  Interventions: Behavioral: PennFit mobile individual intervention
- Online network intervention (Experimental): Behavioral: PennFit mobile online network intervention. Participants were given a Fitbit (zip) to track their daily exercises. Participants used the PennFit app to track their exercises. Participants also received system-generated notifications that reminded them to wear their Fitbit in the morning and to log their activity minutes in the evening. Participants were randomly assigned to 4-person online networks in the PennFit app. Participants in the online networks could see both their own information and the profiles and activity logs of the three other people assigned to their network. In addition, they could send messages to the network through an instant chatting tool.
  Interventions: Behavioral: PennFit mobile online network intervention

INTERVENTIONS:
Behavioral: PennFit mobile individual intervention — PennFit (individual) is a mobile app intervention. Participants received a Fitbit physical activity tracking device and an introductory physical activity promotion session emphasizing the health benefits of physical activity and building skills for daily exercises. Participants used the PennFit app (individual) to record and monitor their own physical activity progress.
  Arms: Individual intervention
Behavioral: PennFit mobile online network intervention — PennFit (online network) is a mobile app intervention. Participants received a Fitbit physical activity tracking device and an introductory physical activity promotion session emphasizing the health benefits of physical activity and building skills for daily exercises. Participants used the PennFit app (online network) to record and monitor their own physical activity progress. They could see both their own information and the profiles and activity logs of the three other women assigned to their network. In addition, they could send messages to the network through an instant chatting tool.
  Arms: Online network intervention

SUMMARY:
Despite the racial disparities in rates of chronic diseases and behaviors linked to chronic diseases, there have been relatively few RCTs of interventions to increase physical activity in African American women. Although some studies found significant improvement on physical activity, most focused on individuals and did not take into consideration the social contexts in which the participants' behaviors occurred. Understanding how online social networks facilitate behavior change can bridge important gaps in the way technology can be used to intervene on health among underserved populations. The primary objective of this study was to test the efficacy of a mobile app (PennFit) intervention in increasing participants' daily active minutes objectively recorded by a fitness tracking device (Fitbit zip). In the control group, participants used the PennFit app to record and monitor their own physical activity progress. In the online social network intervention, participants were randomized to 4-women networks and were able to see and compare their own recorded physical activities with activities of the other three women in their network. Participants in a network had access to an online chatting tool to chat with one another. The secondary objective was to understand the intervention's mechanisms through mediation analysis on theoretical variables.

DETAILED DESCRIPTION:
Despite the racial disparities in rates of chronic diseases and behaviors linked to chronic diseases, there have been relatively few RCTs of interventions to increase physical activity in African American women. Although some studies found significant improvement on physical activity, most focused on individuals and did not take into consideration the social contexts in which the participants' behaviors occurred. A review of qualitative studies of physical-activity correlates in African American adults found that both men and women said group participation would increase their motivation to exercise, and women said that having a physically active partner or friend would facilitate their initiation and maintenance of a physical-activity program. For instance, focus groups with African American women suggested that having a friend or group to exercise with was motivating and should be considered to be an important component of physical activity programs.This finding is consistent with other studies identifying social support as encouraging African American women to engage in physical activity. While previous research emphasized the effects of social support on facilitating physical activity, it is also possible that a lack of social network members perceiving physical activity as a normative behavior may contribute to low rates of physical activity in African American women. Two correlational research found that social support and descriptive norms both predicted physical activity independently . Two experiments found that manipulating descriptive norms increased physical activity . The findings suggest creating physical activity as a normative behavior within African American women's social networks may be an effective way to establish, potentially sustaining physical activity in the long term.

Young African Americans are heavy users of social networking technologies. In 2013, 96% of African Americans aged 18 to 29 used a social networking site of some kind. Understanding how online social networks facilitate behavior change can bridge important gaps in the way technology can be used to intervene on health among underserved populations. The primary objective of this study was to test the efficacy of a mobile app (PennFit) intervention in increasing participants' daily active minutes objectively recorded by a fitness tracking device (Fitbit zip). In the control group, participants used the PennFit app to record and monitor their own physical activity progress. In the online social network intervention, participants were randomized to 4-women networks and were able to see and compare their own recorded physical activities with activities of the other three women in their network. Participants in a network had access to an online chatting tool to chat with one another. The secondary objective was to understand the intervention's mechanisms through mediation analysis on theoretical variables.

ELIGIBILITY:
Inclusion Criteria:

* African American women (self-identified)
* Aged 18 to 35
* Using an Android smartphone
* Residing in Philadelphia

Exclusion Criteria:

* Already participating in another physical activity study
* Not able or willing to carry an Android smartphone
* Being pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Daily active exercise minutes | Intervention day 1 to day 90
  Daily active exercise minutes are recorded by the Fitbit (zip) tracking device

SECONDARY OUTCOMES:
Daily steps | Intervention day 1 to day 90
  Daily steps are recorded by the Fitbit (zip) tracking device
Daily active calories | Intervention day 1 to day 90
  Daily active calories are recorded by the Fitbit (zip) tracking device
Self-reported physical activity | Past 7 days
  The number of days on which participants reported engaging in 20 minutes of vigorous-intensity activity, 30 minutes of moderate-intensity activity, and strength-building activity, in the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: John B Jemmott, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Brackbill D, Yang S, Centola D. Efficacy and causal mechanism of an online social media intervention to increase physical activity: Results of a randomized controlled trial. Prev Med Rep. 2015 Aug 13;2:651-7. doi: 10.1016/j.pmedr.2015.08.005. eCollection 2015. PMID 26844132
- [Background] Jemmott JB 3rd, Jemmott LS, Ngwane Z, Zhang J, Heeren GA, Icard LD, O'Leary A, Mtose X, Teitelman A, Carty C. Theory-based behavioral intervention increases self-reported physical activity in South African men: a cluster-randomized controlled trial. Prev Med. 2014 Jul;64:114-20. doi: 10.1016/j.ypmed.2014.04.012. Epub 2014 Apr 13. PMID 24736094
- [Derived] Zhang J, Jemmott Iii JB. Mobile App-Based Small-Group Physical Activity Intervention for Young African American Women: a Pilot Randomized Controlled Trial. Prev Sci. 2019 Aug;20(6):863-872. doi: 10.1007/s11121-019-01006-4. PMID 30788692